CLINICAL TRIAL: NCT03097874
Title: Confirming the Efficacy/Mechanism of an Adaptive Treatment for Adolescent Anorexia
Brief Title: Adaptive Treatment for Adolescent Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James Dale Lock, MD, PhD, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01MH110538 (NIH); SPO 121859 (Other Grant/Funding Number: NIH); 1R01MH110538-01A1 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Eating Disorder; Anorexia; Anorexia Nervosa; Anorexia in Adolescence; Anorexia in Children; Anorexia Nervosa Restricting Type; Anorexia Nervosa, Atypical; Eating Disorders in Adolescence
Keywords: anorexia; anorexia nervosa; eating disorder; weight; eating; weight loss; family based treatment; FBT; family treatment; therapy; Maudsley method
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia; Anorexia Nervosa; Body Weight; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Based Treatment (Experimental): Family Based Treatment of adolescent Anorexia Nervosa
  Interventions: Behavioral: Family Based Treatment
- Family Based Treatment + Intensive Parental Coaching (Experimental): Family Based Treatment plus Intensive Parental Coaching if weight milestones are not met by session 4.
  Interventions: Behavioral: Family Based Treatment + Intensive Parental Coaching

INTERVENTIONS:
Behavioral: Family Based Treatment — Family Based Treatment of adolescent Anorexia Nervosa
  Other Names: Maudsley Method
  Arms: Family Based Treatment
Behavioral: Family Based Treatment + Intensive Parental Coaching — Family Based Treatment of adolescent Anorexia Nervosa plus an Intensive Parental Coaching component.
  Other Names: FBT + IPC
  Arms: Family Based Treatment + Intensive Parental Coaching

SUMMARY:
The investigators are conducting a randomized controlled trial using an adaptive design for adolescents (ages 12-18) with anorexia nervosa to compare standard Family Based Treatment (FBT) to adaptive FBT with an Intensive Parental Coaching (IPC) component. If participants do not reach expected milestones by session 4 of treatment, participants may be randomized to receive additional IPC or continue treatment as usual with regular FBT.

DETAILED DESCRIPTION:
Potential subjects aged 12 to 18 with anorexia nervosa (AN) will be recruited from Stanford University, University of California, San Francisco, other bay-area medical programs and clinics, and online advertisement to the population at large. If participants are deemed eligible, participants will be invited for a baseline interview (about 2 hours in duration) during which the investigators will conduct interviews and collect questionnaire measures. Then, participants and participants' families will begin Family Based Treatment (FBT) with a study therapist at Stanford University or University of California, San Francisco, respectively. All assessments and treatments are conducted through tele-health.

At session 4, if participants have not gained 2.4kg, an indicator of early treatment response, participants and participants' families will be randomized to receive either treatment as usual (FBT) or an adaptive form of FBT, during which families will receive additional Intensive Parental Coaching (IPC). If participants have reached weight milestones (i.e., 2.4kg at session 4), participants will continue FBT as usual.

At 3 months of treatment and end of treatment, the investigators will collect the same measures taken at baseline. The investigators also ask that families participate in 6- and 12-month follow-up, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age and living with participants' families
* meeting DSM-5 criteria for AN (both subtypes) except for the amenorrhea requirement
* medically stable for outpatient treatment according to the recommended thresholds of the American Academy of Pediatrics and the Society of Adolescent Medicine.

Exclusion Criteria:

* associated physical illness that necessitates hospitalization
* psychotic illness, mental retardation, or any other mental illnesses that would prohibit the use of psychotherapy
* current dependence on drugs or alcohol
* physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight
* previous FBT
* currently taking medication for co-morbid disorders that cannot be safely discontinued on a stable dose for less than 2 months
* in the case of patients with current, or a history of sexual or physical abuse by family members, perpetrators of the abuse will be excluded from treatment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Estimated Body Weight (EBW) | following 9 months of treatment
  individual with anorexia nervosa's body weight at end of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lock JD, Le Grange D, Bohon C, Matheson B, Jo B. Who Responds to an Adaptive Intervention for Adolescents With Anorexia Nervosa Being Treated With Family-Based Treatment? Outcomes From a Randomized Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2024 Jun;63(6):605-614. doi: 10.1016/j.jaac.2023.10.012. Epub 2023 Dec 21. PMID 38142046
- [Derived] L'Insalata A, Trainor C, Bohon C, Mondal S, Le Grange D, Lock J. Confirming the Efficacy of an Adaptive Component to Family-Based Treatment for Adolescent Anorexia Nervosa: Study Protocol for a Randomized Controlled Trial. Front Psychiatry. 2020 Feb 12;11:41. doi: 10.3389/fpsyt.2020.00041. eCollection 2020. PMID 32116856

DOCUMENTS (1):
  • Informed Consent Form (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03097874/ICF_000.pdf